CLINICAL TRIAL: NCT03696706
Title: Effects of Photobiomodulation With Simultaneous Use in a Same LED Device (Red and Infrared) on Clinical Aspects in Individuals With Temporomandibular Dysfunction: Clinical, Randomized, Controlled and Blind Trial.
Brief Title: Photobiomodulation With Red and Infrared LED Device for Temporomandibular Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dowglas
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In the placebo group, the same procedures of the LED group will be made, but the device will be turned off. Participants will not know whether they are in the active or placebo group.
  The investigator will not know to which group the participants belong, only the care provider.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LED group (Active Comparator): LED photobiomodulation will be applied at 36 points, bilaterally, in the temporomandibular joint regions, around these joints, and in the regions of the masseter muscles and anterior part of the temporal muscles, three times a week, totaling 6 treatment sessions, in 2 weeks. The LED apparatus is composed of a flexible rectangular plate (10cm/12cm), which adapts to the format of the area to be treated containing 18 red LEDs - 660 nm and 18 infrared LEDs - 850 nm, with a power of 3.5 mW by LED, 4.45 mW/cm2, radiant exposure of 5.35 J/cm2, radiated area of 14.13 cm2, and energy of 75.6 J.
  Interventions: Radiation: LED photobiomodulation
- Placebo group (Placebo Comparator): For the placebo group, all measures described for the LED group will be adopted, however, the equipment will be switched off.
  Interventions: Radiation: Placebo LED photobiomodulation
- Control group (No Intervention): In this group, the participants will only be evaluated. No intervention will take place.

INTERVENTIONS:
Radiation: LED photobiomodulation — LED photobiomodulation will be applied at 36 points, bilaterally, in the temporomandibular joint regions, around these joints, and in the regions of the masseter muscles and anterior part of the temporal muscles, three times a week, totaling 6 treatment sessions, in 2 weeks. The LED apparatus is composed of a flexible rectangular plate (10cm/12cm), which adapts to the format of the area to be treated containing 18 red LEDs - 660 nm and 18 infrared LEDs - 850 nm, with a power of 3.5 mW by LED, 4.45 mW/cm2, radiant exposure of 5.35 J/cm2, radiated area of 14.13 cm2, and energy of 75.6 J.
  Arms: LED group
Radiation: Placebo LED photobiomodulation — In this group, the same procedures as the LED group will be made, but the device will be turned off.
  Arms: Placebo group

SUMMARY:
Temporomandibular Dysfunction - TMD is considered the main cause of orofacial pain of non-dental origin, and a public health problem. Due to their complexity there are already treatments using various forms of therapy. Photobiomodulation using different light sources, in a single or combined form, makes it possible to use it as another therapeutic resource to be explored. The objective of this study will be to evaluate the effects of photobiomodulation with simultaneous use of light emitting diodes (LEDs), red and infrared, on clinical aspects in individuals with TMD. A randomized, controlled and blind clinical trial is proposed, which will involve 33 individuals (n = 11 per group) of both genders, aged 18-45 years in three groups: Group 1 - LED; Group 2 - placebo and Group 3 - control, submitted to 6 nonconsecutive sessions of photobiomodulation totaling 2 weeks of treatment. The Research Diagnostic Criteria for Temporomandibular Disorders - RDC/TMD will be used to determine the TMD and evaluate the participants. Pain will be assessed using the visual analog scale (VAS), mandibular range of motion will be determined with the aid of a digital caliper, and the electrical activity of the masticatory muscles will be verified by electromyography. A mixed plate of 18 red LEDs - 660 nm and 18 infrared LEDs - 850 nm with power of 3.5 mW per LED, 4.45 mW/cm2, radiant exposure of 5,35 J/cm2, irradiated area of 14.13 cm2, and energy of 75.6 J, in the temporomandibular joint (TMJ) region and in the masseter and temporal muscles, bilateral in 6 sessions. Participants from all groups will be reassessed after the first therapeutic intervention, and again at the end, following the same evaluation procedures used initially.

ELIGIBILITY:
Inclusion Criteria:

* Present TMD;
* Complete dentition (except third molars);
* Present mandibular deviation and/or deflection.

Exclusion Criteria:

* Occlusal changes;
* Use of any type of dental prosthesis;
* Current orthodontic or physiotherapeutic treatment;
* Use of any type of medication during the phases of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Fourteen days.
  VAS is an instrument that allows easy measurement of pain intensity, and consists of a straight line 10 cm long, whose extremities have a verbal description (no pain and worse pain already felt, respectively), in which the participants will be asked to perform a perpendicular trait between the two extremes that represents the level of pain he/she presents at that moment. This will be evaluated at baseline, immediately after treatment and at the end of the treatment.

SECONDARY OUTCOMES:
Range of motion | Fourteen days.
  A digital Starrett® caliper will be used to assess mandibular range of motion (in millimeters), that is, measure mouth opening, lateral deviations (right and left) and protrusion. This procedure composes the clinical evaluation of RDC/TMD. This will be evaluated at baseline, immediately after treatment and at the end of the treatment.
Electromyography | Fourteen days.
  The electrical signals of the right and left masseters and anterior temporal muscles will be captured. We will use an EMG System do Brasil® signal conditioning module, with eight channels (module 830 C), using frequency bandpass filter between 20-1000 Hz, common mode rejection index> 120 db. All data will be collected and processed using a 16-bit analog / digital converter (EMG System do Brasil®). This will be evaluated at baseline, immediately after treatment and at the end of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UniNove, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Sousa DFM, Malavazzi TCDS, Deana AM, Horliana ACRT, Fernandes KPS, Bussadori SK, Mesquita-Ferrari RA. Simultaneous red and infrared light-emitting diodes reduced pain in individuals with temporomandibular disorder: a randomized, controlled, double-blind, clinical trial. Lasers Med Sci. 2022 Dec;37(9):3423-3431. doi: 10.1007/s10103-022-03600-5. Epub 2022 Jun 24. PMID 35751005